CLINICAL TRIAL: NCT06157853
Title: A Randomized, Single-Center, Double-Blinded, Controlled Study Evaluating Procedure Pairing of a Post-Procedure Cream Versus a Comparator in Patients Treated With a Radiofrequency Microneedling for Facial Rejuvenation
Brief Title: Evaluating Procedure Pairing of a Post-Procedure Cream Versus a Comparator in Patients Treated With a Radiofrequency Microneedling for Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RVSN-05-222
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-11

CONDITIONS: Photoaging; Wrinkle
Keywords: post-procedure; radiofrequency microneedling
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: Randomized, single-center, double-blinded, controlled.
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomly assigned to one of the following treatment arms: active post-procedure cream versus comparator anhydrous cream. The products will be packaged in the same container and labelled post-procedure cream. Double blinded study, where the investigator, study subject, and other study personnel involved in the evaluation of the efficacy or safety are blinded to treatment during the 14-day randomization study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Post-Procedure Cream (Active Comparator): Dosage Form: reverse emulsion (water in oil) cream containing bioactive ingredients, botanical actives, peptides, and antioxidants.
  Frequency of Dosage: Twice daily (morning and evening). Subjects will be asked to massage 2 to 3 pumps of test material onto face, forehead, under eyes, cheeks, upper lips, chin, nose, and neck.
  Study duration: 14 days. Active Post-Procedure Cream duration 7-days.
  Interventions: Procedure: Radiofrequency Microneedling; Other: Facial Cleanser; Other: Facial Moisturizer; Other: Sunscreen
- Comparator Anhydrous Cream (Other): Dosage Form: anhydrous cream containing peptides, and antioxidants.
  Frequency of Dosage: Twice daily (morning and evening). Subjects will be asked to massage 2 to 3 pumps of test material onto face, forehead, under eyes, cheeks, upper lips, chin, nose, and neck.
  Study duration: 14 days. Comparator Anhydrous Cream duration 7-days.
  Interventions: Procedure: Radiofrequency Microneedling; Other: Facial Cleanser; Other: Facial Moisturizer; Other: Sunscreen

INTERVENTIONS:
Procedure: Radiofrequency Microneedling — A fractional bipolar radiofrequency microneedling device will be performed at Visit 2, after the 7-day washout period. Subjects were numbed 45 minutes prior to RF microneedling with topical numbing Benzocaine 20%/Lidocaine 6%/tetracaine 4%. Bony areas, periorbital, forehead, and chin were treated with 15 watts at a 2 mm needle depth on cycle mode. All subjects received 20 watts at 3 mm depth on cycle mode on soft tissue, neck, and cheeks.
  Other Names: Fractional biopolar radiofrequency microneedling, InMode
Other: Facial Cleanser — Facial cleanser to be used by subjects twice-daily. This product was used during the entire 14-day study (7-day washout period and 7-day post-procedure timeline).
Other: Facial Moisturizer — Bland moisturizer to be used by subjects twice daily during the 7-day washout period. Use 1 to 2 pumps and place all over face and avoid the eye area.
Other: Sunscreen — Bland sunscreen to be used by subjects after cleansing and the facial moisturizer during the 7-day washout period. Bland sunscreen to be used by subjects after cleansing and after the active post-procedure cream and comparator anhydrous cream. Use the provided sunscreen and reapply as needed throughout the day and per recommendation of the FDA, every 2 hours.
  Other Names: Neutrogena Sheer Zinc SPF 50

SUMMARY:
This randomized, single-center, double-blinded, controlled, clinical trial was conducted to investigate the tolerability, safety, and efficacy of a post-procedure cream when used immediately after radiofrequency microneedling and for seven days post-procedure with twice daily application in healthy female subjects ages 35-65 with moderate facial photodamage (Grade II or III) using the Glogau Scale of Photoaging. Furthermore, this clinical trial will compare the active post-procedure cream to a comparator anhydrous cream product often paired with skin rejuvenation procedures.

A total of 11 healthy female subjects completed the study. Six (6) subjects in the active arm and five (5) subjects in the comparator arm.

DETAILED DESCRIPTION:
This randomized, single-center, double-blinded, controlled, clinical trial was conducted to investigate the tolerability, safety, and efficacy of a post-procedure cream when used immediately after radiofrequency microneedling and for seven days post-procedure with twice daily application in healthy female subjects ages 35-65 with moderate facial photodamage (Grade II or III) using the Glogau Scale of Photoaging in improving patient downtime specifically in minimizing tolerability parameters (erythema, edema, dryness, burning, stinging, and itch) to assist in soothing skin after radiofrequency microneedling procedure.

A 7-day washout period is required for all subjects prior to radiofrequency microneedling procedure. Tolerability (investigator and subject) and safety will be assessed through grading at baseline, post-procedure, post-procedure/post-product application, twenty-four (24) hours post-procedure, three days post-procedure, and seven days post-procedure.

Tolerability parameters included erythema, edema, dryness, burning, stinging, and itch. Efficacy evaluation using the Glogau photoaging scale was performed at screening, baseline, and day 7 post-procedure. The Global Aesthetic Improvement Scale (GAIS) was performed at day 7-post procedure. Self-assessment questionnaire and clinical photography will be completed at all timepoints.

A total of 11 subjects completed study participation. Six (6) subjects in the active arm and five (5) subjects in the comparator arm.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects must be between 35-65 years of age.
2. Female subjects of childbearing potential must be willing to use a form of birth control during the study.
3. Subjects with Fitzpatrick I-VI photo skin type.
4. Subjects must have moderate photodamage (Grade II or III) using the Glogau Scale of Photoaging.

6. Subjects interested in Radiofrequency Microneedling treatments. 7. Subjects must have no skin disease in the facial area being evaluated. 8. Subjects must have no known medical conditions that, in the investigator's opinion, may interfere with study participation. 9. Subjects must be wiling to discontinue all active topical facial products and must only use the assigned study products to the face and neck for the duration of the study.

Exclusion Criteria:

1. Subjects being or planning to become pregnant or breastfeeding during the study
2. Having received a chemical peel, dermabrasion or microneedling treatment in the previous six months; laser resurfacing (ablative, non-ablative) in the previous twelve months
3. Unwilling to refrain from pain medications post-procedure
4. Unwilling to discontinue topical anti-aging facial products for one week prior to study commencement or on prescription strength retinoids or skin lightening produces within two months of the study.
5. Subjects who have a Glogau Score of I or IV.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Investigator Tolerability Scores | 14 days
  The primary tolerability endpoint will be Investigator Tolerability Assessment of erythema, edema, and dryness. A change in scores or lack of significant change after procedure, immediately post-procedure, post product application, Day 1 (24 hours), Day 3, and Day 7 in comparison to baseline (post-procedure) indicates tolerability / safety of the test material. Four-point scale with a lower score indicating a better outcome.
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe
Incidence of Adverse Events | 14-days
  The primary safety endpoint will be determined by the incidence and severity of adverse events in healthy subjects, including immediate post-procedure and through-out the length of the study.
Subject Tolerability Scores | 14 days
  Subject tolerability endpoint will be Subject Tolerability Assessment of burning, itching, and stinging. A change in scores or lack of significant change after procedure, immediately post-procedure, post product application, Day 1 (24 hours), Day 3, and Day 7 in comparison to baseline (post-procedure) indicates tolerability / safety of the test material. Four-point scale with a lower score indicating a better outcome.
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe

SECONDARY OUTCOMES:
Clinical Efficacy Grading | 14 days
  To evaluate the efficacy of the neurocosmetic on self-perceived improvement and objective grading. Investigator clinical grading, using the Glogau photoaging scale performed at Visit 1 (screening), Visit 2 (baseline, 7-days post-washout), and Visit 5 (14 days).
  The Global Aesthetic Improvement Scale (GAIS) to be completed at Visit 5 (14 days).
  GAIS Scoring:
  Very much improved- Optimal cosmetic result for the treatment in this patient. Much improved- Marked improvement in appearance but not completely optimal for this patient. A touch-up would slightly improve the result.
  Improved - Obvious improvement in appearance from the initial condition, but a touch-up or re-treatment is indicated.
  No change- The appearance is the same as than the original condition. Worse- The appearance is worse than the original condition.
Self-Assessment Questionnaire | 14 days
  The secondary efficacy endpoint will be the Self-Assessment Questionnaire. A change in response values at post-procedure/post-product application (Visit 2), Day 1 (Visit 3), Day 3 (Visit 4), and Day 7 (Visit 5) indicates, and improvement compared to baseline response values. Baseline responses will be set to post-procedure/post-product application. Subjects are asked to rate based on a scoring system of the following: from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement / question being asked.

CONTACTS AND LOCATIONS:
Overall Officials: Micahel Gold, MD, Principal Investigator — Tennesse Clinical Research Center
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States